CLINICAL TRIAL: NCT02300519
Title: Thrombin Generation Numerical Models Validation in Haemophilic Case
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Pfizer (Industry); Saint Etienne School of Mine (Other)
Responsible Party: Sponsor
Other Study IDs: 1408185; 2014-A01734-43 (Other: ANSM - FRANCE)
Record Dates: First submitted 2014-11-18; First posted 2014-11-25 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Haemophilia B; Haemophilia A
Keywords: Haemophilia; numerical models; thrombin generation; volunteers; endogenous thrombin potential
MeSH Terms: conditions — Hemophilia B; Hemophilia A | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Volunteers: Blood sampling : 1 blood punction of 36.5 ml for each volunteer
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — Samplings will be taken on 4 citrated S-monovette tubes, 3 citrated tubes and 1 EDTA tube, namely 36.5 ml for each volunteer

SUMMARY:
Personalized therapy in haemophilia has not been reached yet. Treatment is substitutive and its doses are only based on the levels of deficient factor VIII (for haemophilia A) or IX (for haemophilia B). The bleeding severity is not only related to the factor deficiency but also to levels of other coagulation factors (e.g. factor X, II, AT or TFPI). It's necessary to take them into account in order to individualize treatments; and Thrombin Generation Assay (TGA) with the CAT method (Calibrated Automated Thrombography) is a good way because it measures the result of the coagulation cascade. TGA on Platelet Rich Plasma (PRP) is even closer to physiological conditions than on Platelet Poor Plasma (PPP) because platelet influence is represented. It has already been shown (at least in PPP) that the bleeding tendency in haemophilic patients is usually well correlated to TG. Some TG parameters are used to characterize the individual coagulation phenotype, the most important being the Endogenous Thrombin Potential (ETP) and the Lag Time (LT). A hemorrhagic profile usually provides a longer lag time and / or a lower ETP. However, only few studies tried to determine the influence of each coagulation factor and inhibitor on TG. They were done on Platelet Poor Plasma (PPP) or on lyophilized plasma. So the relation between coagulation factors and the different TG parameters remains to be determined, especially in the haemophilic case. It is possible, experimentally, to find the optimal dose of the factor to be added by measuring TG in samples with different factor VIII or IX concentrations, but this method would be time consuming and expensive, especially because it should be done for each haemophilic patient. A better way consists in using TG numerical models. For a set of initial factor levels they simulate the TG and its associated parameters. It is now essential to validate the existing models, especially in haemophilic cases, in order to see whether they are reliable and can be used in clinical practice afterwards.The objective of this study is to validate thrombin generation numerical models which could predict the factor VIII or IX activity correction to reach a thrombin generation sufficient to avoid bleeding. A comparison between the TG observed in haemophilic patients and the TG predicted by the models is needed to validate the models. In order to define a 'safe' TG i.e. sufficient to avoid bleeding, normal ranges of TG parameters have to be measured.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form
* Age between 18 and 45 years old
* Male
* no smoker

Exclusion Criteria:

* other clinical research protocol participation during the 3 months before inclusion
* Personal or familial history of hemorrhagic disease (parents, brothers and sisters
* Personal history of thrombosis (arterial or venous)
* Familial history of thrombosis before 45 years old (parents, brothers and sisters)
* Drug treatments of aspirin or anti-inflammatory type during the week before sampling
* Surgery the month before sampling
* Chronic pathology responsible for inflammatory syndrome
* Infectious episode in course

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: volunteers witch work in CHU Saint-Etienne
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Endogenous Thrombin Potential (ETP) predicted by numerical models | up to 12 monthes
  ETP (i.e. the aera under the thrombin generation curve, nM.min) measured in haemophilic patients is compared to ETP predicted by numerical models.
Lag Time of the thrombin generation curve predicted by numerical models | up to 12 monthes
  Lag time (min) measured in haemophilic patients is compared to the lag time predicted by numerical models
Peak value of the thrombin generation curve predicted by numerical models | up to 12 monthes
  Peak value (nmol thrombin) measured in haemophilic patients is compared to the peak value predicted by numerical models
Time to peak (TTP) of the thrombin generation curve predicted by numerical models | up to 12 monthes
  TTP (min) measured in haemophilic patients is compared to TTP predicted by numerical models
Velocity Index (V) of the thrombin generation curve predicted by numerical models | up to 12 monthes
  Velocity Index measured in haemophilic patients is compared to TTP predicted by numerical models

SECONDARY OUTCOMES:
Endogenous Thrombin Potential (ETP) for volunteers | day 1
  ETP (i.e. the aera under the thrombin generation curve, nM.min) is measured by Thromboplastin Generation Tests (TGTs)
Lag Time of the thrombin generation curve for volunteers | day 1
  Lag time (min) of the thrombin generation curve is measured by Thromboplastin Generation Tests (TGTs)
Peak value of the thrombin generation curve for volunteers | day 1
  Peak value of the thrombin generation curve is measured by Thromboplastin Generation Tests (TGTs)
Time to peak (TTP) of the thrombin generation curve for volunteers | day 1
  TTP of the thrombin generation curve is measured by Thromboplastin Generation Tests (TGTs)
Velocity Index (V) of the thrombin generation curve for volunteers | day 1
  Velocity Index (V) of the thrombin generation curves measured by Thromboplastin Generation Tests (TGTs)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte TARDY-PONCET, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France